CLINICAL TRIAL: NCT02986152
Title: Cancer Distress Coach Mobile App Randomized Controlled Trial
Brief Title: Cancer Distress Coach Mobile App Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Institute for Health Innovation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00075411
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Posttraumatic Stress Disorder; Cancer
Keywords: PTSD; anxiety; depression; distress; fear; coping; support; caregiver; oncology; app; mobile app
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Neoplasms; Anxiety Disorders; Depression; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDC Mobile App Treatment (Experimental): Subjects who are randomized to the CDC mobile app treatment arm will be asked to perform the app's full suite of intervention tools such as learning about PTSD, assessment, finding support, and mind/body exercises (e.g., guided imagery, meditation, and relaxation exercises) over the entire 8-week study period.
  Interventions: Behavioral: Cancer Distress Coach Mobile App
- CDC Mobile App Wait-List Control (Other): Subjects who are randomized to the CDC mobile app wait-list control arm will be asked to perform only the learning about PTSD, assessment, and finding support activities for the first 4 weeks. Following completion of the Week-4 questionnaires, subjects will then be asked to additionally perform the mind/body exercises (e.g., guided imagery, meditation, and relaxation exercises) for the duration of the 8-week study period.
  Interventions: Behavioral: Cancer Distress Coach Mobile App

INTERVENTIONS:
Behavioral: Cancer Distress Coach Mobile App — Cancer Distress Coach is a stand-alone symptom management tool with three basic components. The Learn about Distress module provides psycho-education. The Insights module includes an inspiring Quote of the Day, daily activity planning tips, a graph displaying the user's distress level plotted over time, and assessment feedback. The main action of the application is in the Activities module that provides patients with skills to manage their stress in the moment they experience it. Depending on the severity, the patient is routed to any of a number of helpful skills based on cognitive-behavioral principles. The stress management tools include positive imageries, soothing songs and pictures, and the Relax-Identify-Decide tool. Also included is "find support" and "get support now" to connect the user to his/her support network and locate informal cancer and non-cancer related support or (immediate) professional care.
  Other Names: CDC Mobile App

SUMMARY:
The Cancer Distress Coach (CDC) mobile app is a symptom management tool for posttraumatic stress disorder (PTSD) in cancer patients and caregivers. Based largely on "PTSD Coach" from the National Center for PTSD, the CDC app was redesigned for both iOS and Android platforms and is tailored specifically to individuals impacted by cancer.

This study aims to evaluate whether CDC app usage influences symptoms of PTSD through a randomized controlled trial (RCT) where subjects are placed into either the intervention group or the wait-listed control group for a period of 8 weeks. The CDC app is available as a free download on the App Store® and on Google Play™.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with cancer or are/were a caregiver to someone with cancer
* Resident of the United States of America
* Able to read and write English
* Age ≥ 18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-04-13 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms as measured by the PTSD Checklist (PCL-5) | Baseline, Week 4, Week 8
  The PCL-5 is a 20-item self-report symptom checklist that closely mirrors DSM-5 diagnoses criteria. The instructions will be modified so that symptoms are keyed to the particular traumatic stressor of interest; specifically, subjects will be asked to rate each PTSD symptom in the past 4 weeks with respect to their cancer diagnosis and treatment.

SECONDARY OUTCOMES:
Change in distress level as measured by the Distress Thermometer | Baseline, Week 4, Week 8
  The Distress Thermometer is used to assess psychosocial distress. It consists of a one-item self-report scale from 0-10, where 0 represents no distress and 10 represents extreme distress.
Change in stress management self-efficacy as measured by the Self-efficacy questionnaire | Baseline, Week 4, Week 8
  The Self-efficacy questionnaire is a 1-item measure of self-efficacy developed by the National Center for PTSD. It rates one's ability to manage the stress of situations reminiscent of the cancer experience on a scale of 0-4, where 0 is not at all able and 4 is extremely able.

OTHER OUTCOMES:
Feasibility as measured by satisfaction with the Cancer Distress Coach mobile app, as measured by the Feedback questionnaire | Week 4, Week 8
  The Feedback questionnaire was developed by the study team to assess perceived helpfulness of the app and user satisfaction with the app. Points are totaled and summed.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia K Smith, PhD, MSW, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No